CLINICAL TRIAL: NCT01606241
Title: A Phase I Trial of the Safety and Immunogenicity of a Multi-epitope Folate Receptor Alpha Peptide Vaccine Used in Combination With Cyclophosphamide in Subjects Previously Treated for Breast or Ovarian Cancer
Brief Title: Vaccine Therapy and Cyclophosphamide in Treating Patients With Stage II-III Breast or Stage II-IV Ovarian, Primary Peritoneal, or Fallopian Tube Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MC1015; NCI-2012-00586 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); MC1015 (Other: Mayo Clinic)
Record Dates: First submitted 2012-05-23; First posted 2012-05-25 (Estimated); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Recurrent Breast Carcinoma; Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma; Stage IIA Breast Cancer; Stage IIA Fallopian Tube Cancer; Stage IIA Ovarian Cancer; Stage IIB Breast Cancer; Stage IIB Fallopian Tube Cancer; Stage IIB Ovarian Cancer; Stage IIC Fallopian Tube Cancer; Stage IIC Ovarian Cancer; Stage IIIA Breast Cancer; Stage IIIA Fallopian Tube Cancer; Stage IIIA Ovarian Cancer; Stage IIIA Primary Peritoneal Cancer; Stage IIIB Breast Cancer; Stage IIIB Fallopian Tube Cancer; Stage IIIB Ovarian Cancer; Stage IIIB Primary Peritoneal Cancer; Stage IIIC Breast Cancer; Stage IIIC Fallopian Tube Cancer; Stage IIIC Ovarian Cancer; Stage IIIC Primary Peritoneal Cancer; Stage IV Fallopian Tube Cancer; Stage IV Ovarian Cancer; Stage IV Primary Peritoneal Cancer
MeSH Terms: conditions — Breast Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — Cyclophosphamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (cyclophosphamide and vaccine therapy) (Experimental): Patients receive cyclophosphamide PO BID on days 1-7 and 15-21 of course 1. Within 3-5 days, patients receive multi-epitope folate receptor alpha peptide vaccine ID on day 1. Vaccine treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cyclophosphamide; Other: Laboratory Biomarker Analysis; Biological: Multi-epitope Folate Receptor Alpha Peptide Vaccine

INTERVENTIONS:
Drug: Cyclophosphamide — Given PO
  Other Names: (-)-Cyclophosphamide; 2H-1,3,2-Oxazaphosphorine, 2-[bis(2-chloroethyl)amino]tetrahydro-, 2-oxide, monohydrate; Carloxan; Ciclofosfamida; Ciclofosfamide; Cicloxal; Clafen; Claphene; CP monohydrate; CTX; CYCLO-cell; Cycloblastin; Cycloblastine; Cyclophospham; Cyclophosphamid monohydrate; Cyclophosphamidum; Cyclophosphan; Cyclophosphane; Cyclophosphanum; Cyclostin; Cyclostine; Cytophosphan; Cytophosphane; Cytoxan; Fosfaseron; Genoxal; Genuxal; Ledoxina; Mitoxan; Neosar; Revimmune; Syklofosfamid; WR- 138719
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Multi-epitope Folate Receptor Alpha Peptide Vaccine — Given ID
  Other Names: FR Alpha Peptide Vaccine

SUMMARY:
This phase I clinical trial studies the side effects of vaccine therapy and cyclophosphamide in treating patients with stage II-III breast cancer or stage II-IV ovarian, primary peritoneal or fallopian tube cancer. Vaccines made from peptides may help the body build an effective immune response to kill tumor cells. Drugs used in chemotherapy, such as cyclophosphamide, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Giving vaccine therapy and cyclophosphamide may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the safety of administering one cycle of cyclophosphamide and six subsequent monthly vaccinations with a peptide-based vaccine targeting folate receptor (FR)-alpha (multi-epitope folate receptor alpha peptide vaccine).

II. To assess the ability of this vaccination protocol to elicit an immune response as measured by activated FR-alpha-specific T lymphocytes or high-affinity antibodies.

SECONDARY OBJECTIVES:

I. To determine FR-alpha expression status of primary tumors when available as formalin-fixed, paraffin-embedded material and whether expression correlates with the ability to generate an immune response.

II. To identify human lymphocyte antigen (HLA) class I binding peptides from FR-alpha that are recognized by lymphocytes from patients prior to and after vaccination.

III. To determine whether cyclophosphamide treatment, prior to vaccination, results in regulatory T cell depletion by assessing regulatory T cells before and immediately after cyclophosphamide treatment.

IV. To compare FR-alpha (FRa) expression levels in tumor removed at primary surgery to FRa expression levels in tumor removed for clinical purposes at disease recurrence. (For ovarian cancer patients whose disease recurs.)

OUTLINE:

Patients receive cyclophosphamide orally (PO) twice daily (BID) on days 1-7 and 15-21 of course 1. Within 3-5 days, patients receive multi-epitope folate receptor alpha peptide vaccine intradermally (ID) on day 1. Vaccine treatment repeats every 28 days for up to 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3, 6, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Clinically confirmed no evidence of disease >= 90 days from completion of systemic therapy with the exception of hormonal therapy and bisphosphonates (per practice guidelines for breast and ovarian cancer)
* Histological or cytological confirmation of stage II or III breast cancer or stage II, III, or IV ovarian/primary peritoneal/fallopian tube cancer; Note: patients with stage IV ovarian/primary peritoneal/fallopian tube cancer must register within one year of completing chemotherapy
* Completed systemic treatment (chemotherapy, immune modulators [such as trastuzumab], radiation, and/or corticosteroids) with the exception of hormonal therapy and bisphosphonates >= 90 days prior to registration
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0 or 1
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelets >= 100,000/ul
* Hemoglobin >= 10.0 g/dL
* Creatinine =< 1.5 x upper limit of normal (ULN) or 24 hour urine =< grade 2
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) =< 3 x ULN
* Serum albumin >= 3 g/dL
* Urinalysis with =< 2+ proteinuria
* Thyroid-stimulating hormone (TSH) - negative or =< normal institutional range
* Anti-nuclear antibody (ANA) - negative or =< normal institutional range
* Serum rheumatoid factor (RF) - negative or =< normal institutional range
* Negative serum pregnancy test done =< 7 days prior to registration, for women of childbearing potential only
* Capable of understanding the investigative nature, potential risks, and benefits of the study and capable of providing valid informed consent
* Willing to return to Mayo Clinic Rochester for follow-ups (immunizations, blood draws, etc.)
* Willing to provide mandatory blood samples for primary and correlative goals
* Willing to receive a tetanus vaccination if you have not had one within the past year

Exclusion Criteria:

* Any of the following:

  * Pregnant women
  * Nursing women unwilling to stop breast feeding
  * Men or women of childbearing potential who are unwilling to employ adequate contraception from the time of registration through cycle 6 (or the final vaccine cycle for each patient)
* Co-morbid systemic illnesses or other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study or interfere significantly with the proper assessment of safety and toxicity of the prescribed regimens
* Immunocompromised patients (other than that related to the use of corticosteroids) including patients known to be human immunodeficiency virus (HIV) positive
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Receiving any other investigational agent
* Other active malignancy =< 5 years prior to registration; EXCEPTIONS: Non-melanoma skin cancer or carcinoma-in-situ of the cervix; NOTE: If there is a history of prior malignancy, they must not be receiving other specific treatment (cytotoxics, monoclonal antibodies, small molecule inhibitors) for this cancer
* Known history of autoimmune disease
* Any contraindication to receiving sargramostim (GM-CSF) or cyclophosphamide
* Uncontrolled acute or chronic medical conditions including, but not limited to the following:

  * Active infection requiring antibiotics
  * Congestive heart failure (New York Heart Association class III or IV; moderate to severe objective evidence of cardiovascular disease)
  * Myocardial infarction or stroke within previous 6 months
* Use of a systemic steroid =< 30 days prior to registration
* Receiving thyroid replacement therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2012-07-24 (Actual); Primary Completion 2014-09-25 (Actual); Study Completion 2018-03-09 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who experience severe toxicities (grades 3-5 of the National Cancer Institute's Cancer Therapy Evaluation Program [CTEP] Common Terminology Criteria for Adverse Events, version 4.0) | Up to 12 months
  Defined as adverse events that are classified as either unrelated, unlikely to be related, possibly, probably, or definitely related to study treatment. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed by primary disease site to determine toxicity patterns.

SECONDARY OUTCOMES:
Disease-free survival | Time from registration to documentation of disease recurrence, second primary, or death without disease recurrence or second primary, assessed up to 12 months
  The distribution of disease-free survival will be estimated using the method of Kaplan-Meier for each disease group (breast cancer; ovarian cancer).
FRa expression | Up to 12 months
  A 90% binomial confidence interval will be constructed for percentage of patients who develop an immune response among those patients who have FRa positive disease. Similarly, a 90% binomial confidence interval will be constructed for percentage of patients who develop an immune response among those patients who have FRa negative disease.
Overall survival time | Time from registration to death due to any cause, assessed up to 12 months
  The distribution of overall survival times will be estimated using the method of Kaplan-Meier for each disease group (breast cancer; ovarian cancer).
Percentage change in plasma concentration of cytokines and chemokines | Baseline to up to 12 months
  The percent change in plasma concentrations of cytokines and chemokines from pre-treatment concentrations will be determined. Will be plotted against time with the points belonging to a particular individual connected. Each graph will be visually inspected for trends across time and difference between treatment regimens.

OTHER OUTCOMES:
FR-alpha -specific antibody response by enzyme linked immunosorbent assay | Up to 12 months
  A vaccine-induced FR-alpha-specific antibody responses will be defined as (1) a 2-fold or greater increase in FR-alpha-specific antibody concentration from pretreatment levels at any point during treatment or (2) FR-alpha-specific antibodies above the lower limit of detection at any point during treatment if pre-treatment levels were non-detectable.
FR-alpha-specific antibody response by enzyme-linked immunospot | Up to 12 months
  A patient is said to have an antigen-specific response at a given post-treatment time point if one of the following sets of conditions is true: 1) the average antigen specific value at pre-treatment > 0, there is a 2 fold increase in average antigen-specific value at post treatment time relative to antigen specific value at pretreatment, and the post-treatment time point of interest (INT) is wholly above the pre-INT; or (2) the average antigen specific value at pre-treatment =< 0, the average antigen-specific value at post treatment time > 0, and the post-INT is wholly above the pre-INT.
Percent change in antigen-specific cytokine profiles | Baseline to up to 12 months
  Percent change in plasma concentrations of cytokines from pre-treatment levels will be examined to determine skewing of the T cell response to type 1 helper cell or type 2 helper cell after vaccination.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew S. Block, M.D., Ph.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States